CLINICAL TRIAL: NCT01520467
Title: Efficacy and Tolerance of Treatment With an Aromatase Inhibitor (Anastrozole) to Limit the Progression of Bone Maturation Related to Pathological Adrenarche in Children With Silver-Russell or Prader-Willi Syndrome
Brief Title: Aromatase Inhibitor in Bone Maturation, Children With Silver Russell or Prader-Willi Syndrome
Acronym: ANASILPRA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P 100129; AOM 10093 (Other: Assistance Publique)
Record Dates: First submitted 2012-01-25; First posted 2012-01-30 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Silver Russell Syndrome; Prader-Willi Syndrome
Keywords: SRS; PWS; pathological adrenarche; aromatase inhibitor; Children
MeSH Terms: conditions — Silver-Russell Syndrome; Prader-Willi Syndrome | interventions — Anastrozole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anastrozole (Experimental): stratification according to the rare disease. Oral administration of Anastrozole (1mg/day) for 18 months
  Interventions: Drug: Anastrozole
- Placebo (Placebo Comparator): stratification according to the rare disease. Oral administration of 1 placebo tablet /day for 18 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anastrozole — Anastrozole (1mg/day), administered orally for 18 months
  Arms: Anastrozole
Drug: Placebo — 1 placebo tablet /day administered orally for 18 months.
  Arms: Placebo

SUMMARY:
There is currently no drug with pediatric marketing authorization capable of limiting the advance in bone maturation of children with aggressive adrenarche. Estrogens are the principal actors involved in bone maturation and premature epiphyseal fusion. Aromatase inhibitors, used for the treatment of hormone-dependent cancers, block the transformation of androgens into estrogens. Third generation inhibitors, of which Anastrozole is one, appear to be well tolerated in children and are sometimes used within the framework of clinical trials to limit bone maturation and improve prognosis with respect to final size, notably in children treated with growth hormone (GH) due to a GH deficit. Nevertheless, the data reported are based on small sample sizes and do not include children with pathological adrenarche.

DETAILED DESCRIPTION:
Silver-Russell syndrome (SRS), which occurs secondary to an imprinting disorder due to the anomalous methylation of chromosome 11 or due to a uniparental disomy of chromosome 7, is a rare syndrome (ORPHA813, OMIM 180860) characterized by growth retardation with an intrauterine onset, a normal head circumference, small postnatal size and major feeding difficulties. Starting at a very young age, the rapid aging of bone can occur even in the absence of central puberty, in association with the production of androgens by the adrenal glands (adrenarche). This advanced bone maturation can compromise final size, even when the child receives growth hormone (GH) treatment for several years.

Prader-Willi syndrome (PWS) is also a rare disease (ORPHA739, OMIM 176270), occurring secondary to an imprinting disorder due to an anomaly in chromosome 15 (paternal deletion or maternal disomy). These children also present feeding difficulties during the first few years of life, as well as small size. They are frequently treated with GH, and their bone age can increase during the course of adrenarche, as in certain patients with SRS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with genetically proven SRS or PWS, under treatment with GH in the usual context of the disease, presenting with adrenarche (defined either by DHEAS levels as a function of age or by the appearance of pubic hair) associated with a bone age at least 6 months greater than chronological age and in the absence of the onset of central puberty (LH peak ≤ LH peak in prepubertal patients, according to the standards of the laboratory performing the GnRH stimulation test for LH and FSH, and dating back to less than 3 months).
* Patients with medical coverage.
* The lower age limit for inclusion is 5 years and the upper age limit is 10 complete years for girls and 12 complete years for boys.
* The maximum body-mass index (BMI) Z-score for inclusion is +4
* Patients should be capable of swallowing pills of the same size as the experimental drug.

Exclusion Criteria:

* Renal insufficiency (creatinine clearance, calculated according to the Schwartz formula, lower than 70ml/min/l, 73 m²),
* Hepatic insufficiency (prothrombin ratio < 50% and factor V < 50%),
* Hepatic cytolysis (liver transaminases levels greater than twice the normal level for age), cholestasis (gamma-glutamyl transferase (GGT) levels greater than twice the normal level for age),
* Contraindication to one of the components of Anastrozole or the placebo.
* Patients with scoliosis requiring surgery.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2012-04; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
The rate of success in each of the two groups, evaluated using an X-ray of the left hand and wrist. Success is defined as a difference in the rate of progression of bone maturation of at least 9 months after 18 months of treatment. | 18 months
  Principal objective: To evaluate the efficacy of Anastrozole compared to placebo in slowing bone maturation during pathological adrenarche in children with SRS or PWS.
  Principal criterion of evaluation: The rate of success in each of the two groups, evaluated using an X-ray of the left hand and wrist. Success is defined as a difference in the rate of progression of bone maturation of at least 9 months after 18 months of treatment.

SECONDARY OUTCOMES:
metabolic impact (monitoring of body composition by bi photonic absorptiometry, lipid, glucose, HbA1c, insulin and HOMA-IR profiles, leptin). | baseline, 6, 12 and 18 months
impact on bone (X-ray of the dorsolumbar spine, bi photonic absorptiometry, blood-borne markers of bone remodeling). | 18 months, and earlier in case of bone pain
impact on the gonadotropic axis | baseline, 6, 12 and 18 months
impact on the somatotropic axis (growth rate, IGF-1, IGFBP3). | baseline, 6, 12 and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Irène Netchine, MD, PhD, Principal Investigator — Assistance Publique
Locations (1):
- Explorations Fonctionnelles d'Endocrinologie - Centre de Référence des Maladies Endocriniennes Rares de la Croissance Hôpital Armand Trousseau, Paris, France